CLINICAL TRIAL: NCT07146373
Title: The Effect of Strengthening Respiratory Muscles on Cognitive and Physical Functioning in Patients With Neurocognitive Disorders
Brief Title: Effect of Inspiratory Muscle Training in Cognition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, IRINI PATSAKI, Assistant Professor, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 27134
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: mild cognitive impairement; dementia; respiratory physiotherapy; inspiratory muscle training
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (Experimental): IMT that consists of 5set/6 breaths at 50-60% of Maximal Inspiratory Pressure, 5 session per weak for 3 months.
  Physical and Cognitive training
  Interventions: Other: Inspiratoty Muscle training
- Control (Active Comparator): Physical and cognitive training
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Inspiratoty Muscle training — Participants will follow an IMT program through a threshold IMT device which consists of 5 set/6 breaths at 50-60% MIP for 3 months along with their usual physical and cogntive training
  Arms: Inspiratory Muscle Training
Other: Usual Care — Physical and cognitive training
  Arms: Control

SUMMARY:
The goal of this clinical trial is to examine the effect of a respiratory muscle strengthening program on the cognitive and physical functioning of patients with neurocognitive disorders (Mild Cognitive Impairment) or those predisposed to them.

The main questions that aims to answer are:

1. Is Inpsiratory Muscle Training (IMT) feasible in people with mild cognitive impairement?
2. Could Inspiratory Muscle Training (IMT) improve congitive function in people with mild cognitive impairement?
3. Could Inspiratory Musclre training improve physical function in this population?

Participants will be:

1. < 60 age or > 90 age
2. MMSE (Mini Mental State Examination) score ≤ 28 and ≥ 18 and follow a high intensity IMT program along with a physical - cognitive program. or just the physical - cognitive program.

ELIGIBILITY:
Inclusion Criteria:

* MMSE (Mini Mental State Examination) score ≤ 28 και ≥ 18
* stable treatment related to medication

Exclusion Criteria:

* MMSE score < 18 και > 28
* psychological disorder
* any contraindication to physical training

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination | T0 at the beginning, T1 at 3 months (end of intervention), T2 at 6 months (follow-up)

SECONDARY OUTCOMES:
Frontal Assessment Battery | T0 at the beginning, T1 at 3 months (end of intervention), T2 at 6 months (follow-up)
Addenbrooke's Cognitive Examination | T0 at the beginning, T1 at 3 months (end of intervention), T2 at 6 months (follow-up)
Time up and Go (TUG) | T0 at the beginning, T1 at 3 months (end of intervention), T2 at 6 months (follow-up)
Sit-to-Stand test | T0 at the beginning, T1 at 3 months (end of intervention), T2 at 6 months (follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: IRINI PATSAKI, PhD, Principal Investigator — University of West Attica
Locations (1):
- University of West Attica, Aigáleo, Attica, Greece

IPD SHARING:
Plan to Share IPD: No